Microvascular and anti-inflammatory effects of Rivaroxaban compared to low dose aspirin in type 2 diabetic patients with very high cardiovascular risk and subclinical inflammation (MicroVasc-DIVA)

## **Statistical Analysis Plan (SAP)**

**Primary trial objective:** Evaluation of efficacy defined as the difference of change

of forearm blood flow with venous occlusion

plethysmography at baseline and after forearm ischemia after 20 weeks treatment between rivaroxoban and aspirin

therapy.

Additionally the difference of arterial stiffness after 52 weeks treatment (extension study) between rivaroxoban

and aspirin therapy will be evaluated.

**Trial design:** Multicenter, prospective, active controlled,

randomized, 2 parallel arms, open

interventional clinical trial

Investigational

medicinal product:

Rivaroxaban

**Comparator:** 

Aspirin

Clinical study phase:

Phase IIIb

PD Dr.

Date:

19.09.2018

1.0

**EudraCT No.:** 

**Investigator:** 

2014-001305-41

Version:

**GWT-TUD GmbH** 

**Principal Coordinating** 

Frank Pistrosch

Sponsor:

Dresden -

Germany

Statistician:

Dr. Dorothea Schipp

#### Confidential

The information provided in this document is strictly confidential and is intended solely for the guidance of the clinical investigation. Reproduction or disclosure of this document, whether in part or in full, to parties not associated with the clinical investigation or its use for any other purpose without the prior written consent of the sponsor is not permitted.

This SAP is produced on a word-processing system and bears no signatures.

The approval of the SAP is documented in a separate Signature Document.

### Signatures

| Sponsor: | GWT-TUD GmbH | |
|---|---|---|
| Sponsor. | Freiberger Strasse 33 | |
| | 01067 Dresden/Germany | |
| | Phone: +49 (0) 351 25933 100 Fax: +49 (0) 351 25933 111 E-mail: contact@gwtonline.de | |
| | Signature of Sponsor's Representative | 20, 9, 1P<br>Date |
| | Dr. Carda tobles Printed Name of Representative | |
| | Signature of Principle Coordinating Investigator | Date |
| > | Printed Name of Principle Coordinating Investigator | |
| | Signature of Statistician | 21.9.18<br>Date |
| | Dr. Dorothea Schipp Printed Name of Statistician | - |

## **Signatures**

| GWT-TUD GmbH | |
|----------------------------------------|----------|
| Freiberger Strasse 33 | (4 |
| 01067 Dresden/Germany | |
| and a contracting | |
| Phone: +49 (0) 351 25933 100 | |
| Fax: +49 (0) 351 25933 111 | |
| E-mail: contact@gwtonline.de | |
| 11/ 461/121 | 0 - 0 15 |
| Signature of Spansor's P | 20. 7. 1 |
| Signature of Sponsor's Representative | Date |
| Dr. Corda Kohler | |
| Printed Name of Representative | < 9 |
| The traine of hepresentative | |
| Att | |
| 1/1/ | |
| VVV C | 21.9.18 |
| Signature of Principle Coordinating | Date |
| Investigator | Date |
| PD Or Frank Pistrosch | |
| Printed Name of Principle Coordinating | |
| Investigator | |
| v v | |
| Signature of Statistician | Date |
| | Date |
| Printed Name of Statistician | |

## **Table of Contents**

| Si | gnature | es | | 2 |
|----|---------|---------|-------------------------------------------|----|
| 1 | Rati | onal | of the statistical analysis plan | 6 |
| 2 | Inve | stiga | tional Plan | 6 |
| | 2.1 | Stud | dy design | 6 |
| | 2.2 | Visit | t schedule | 7 |
| | 2.3 | Stud | dy objectives | 8 |
| | 2.3. | 1 | Primary objectives | 8 |
| | 2.3.2 | 2 | Secondary objectives | 9 |
| | 2.3.3 | 3 | Explorative study objective(s) | 9 |
| | 2.4 | Sam | ple size calculation | 9 |
| 3 | Ana | lysis | Sets | 10 |
| | 3.1 | Full | Analysis Set (FAS) | 10 |
| | 3.2 | Safe | ety Analysis Set (SAF) | 10 |
| | 3.3 | Per- | Protocol Set (PPS) | 10 |
| 4 | Ana | lysis ' | Variables | 10 |
| | 4.1 | Den | nographics | 10 |
| | 4.2 | Med | dical history | 10 |
| | 4.3 | Con | comitant medication and acute diseases | 11 |
| | 4.4 | Dru | g administration | 11 |
| | 4.5 | Effic | cacy Variables | 11 |
| | 4.6 | Lab | oratory Variables | 11 |
| | 4.7 | Safe | ety Variables | 12 |
| | 4.7. | 1 | Vital Signs | 12 |
| | 4.7.2 | 2 | Safety laboratory | 12 |
| | 4.7.3 | 3 | Adverse Events and Serious Adverse Events | 12 |
| | 4.8 | Defi | nition of derived variables | 12 |
| | 4.8. | 1 | Primary variable | 12 |
| | 4.8.2 | 2 | Secondary variables | 13 |
| 5 | Effic | acy E | Endpoints | 13 |
| | 5.1 | Prin | nary endpoint | 13 |
| | 5.2 | Seco | ondary endpoints | 13 |
| 6 | Stat | istica | ll Methods | 13 |
| | 6.1 | Data | a Handling | 13 |
| | 6.2 | Des | criptive or summary statistics | 13 |
| | 6.3 | Нур | othesis Testing | 13 |
| | 6.4 | Sub | ject Disposition | 14 |
| | 6.5 | Den | nographics | 14 |

| | 6.6 | Med | dical History | 14 |
|---|------|-------|-----------------------------------------------------|----|
| | 6.7 | Con | comitant medication and Acute Diseases | 15 |
| | 6.8 | Con | npliance | 15 |
| | 6.9 | Trea | atment exposure and observation period | 15 |
| | 6.10 | Ana | lysis of baseline characteristics | 15 |
| | 6.11 | Ana | lysis of Efficacy Endpoints | 15 |
| | 6.11 | 1.1 | Analysis of Primary Endpoint | 15 |
| | 6.11 | 2 | Analysis of Secondary Endpoints | 16 |
| | 6.12 | Ana | lysis of Safety Data | 16 |
| | 6.12 | 2.1 | Vital Signs | 16 |
| | 6.12 | 2.2 | Safety Laboratory Measurements | 16 |
| | 6.12 | 2.3 | Adverse Events | 16 |
| | 6.12 | 2.4 | Bleedings | 17 |
| | 6.13 | Inte | rim analysis | 17 |
| | 6.14 | Rep | orting conventions | 17 |
| 7 | Арр | endix | k: Mock-Up tables, figures and listings | 18 |
| | 7.1 | Sub | jects Disposition | 18 |
| | 7.2 | Den | nographics | 20 |
| | 7.3 | Med | dical History | 21 |
| | 7.3. | 1 | Medical History | 21 |
| | 7.3. | 2 | Concomitant medication | 21 |
| | 7.3. | 3 | ECG and Pregnancy Test | 21 |
| | 7.4 | Con | npliance | 22 |
| | 7.5 | Trea | atment exposure and observation period | 23 |
| | 7.6 | Effic | cacy Endpoints | 24 |
| | 7.6. | 1 | Forearm Blood Flow (FBF) | 24 |
| | 7.6. | 2 | Pulse Wave Analysis | 26 |
| | 7.6. | 3 | Laser Doppler fluxometry (LDF) | 29 |
| | 7.7 | Effic | cacy Laboratory | 30 |
| | 7.7. | 1 | Inflammation Laboratory | 30 |
| | 7.7. | 2 | Laboratory for Endothelian Function and Coagulation | 31 |
| | 7.8 | Safe | ety Variables | 33 |
| | 7.8. | 1 | Vital Signs | 33 |
| | 7.8. | 2 | Safety Laboratory | 35 |
| | 7.8. | 3 | Adverse Events | 36 |
| | 78 | 4 | Bleedings | 36 |

#### **Abbreviations**

**Abbreviation Definition** 

ADR Adverse Drug Reaction

AE Adverse Event

ANCOVA Analysis of Covariance b.i.d. (Bis in Die) twice a day BMI Body Mass Index CI Confidence Interval

CRNM Clinical Relevant Non-Major CSV Clinically significant value

CTCAE Common Terminology Criteria for Adverse Events

ECG Electrocardiogram

eCRF Electronical Case Report Form

FAS Forearm Blood Flow

GmbH Gesellschaft mit beschränkter Haftung ICH International Council for Harmonization

LDF Laser Doppler Fluxometry
LLOQ Lower Limit of Quantification

Max Maximum
Min Minimum
OR Odds Ratio

PCSV Potentially clinically significant value

PPS Per Protocol Set
PT Preferred Term
PWA Pulse Wave Analysis
PWV Pulse Wave Velocity
q.d. (quaque die) daily

SADR Serious Adverse Drug Reaction

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAF Safety Analysis Set
SOC System Organ Class

SOP Standard Operating Procedure

STD Standard Deviation

vs. versus

#### 1 Rational of the statistical analysis plan

The purpose of the statistical analysis plan (SAP) is to ensure the credibility of the study results by prespecifying statistical approaches for the analysis of study. The SAP is intended to be a comprehensive and detailed description of strategy and statistical techniques to be used to realize the analysis of data for the MicroVasc-DIVA study.

This plan may be revised during the study to accommodate protocol amendments and to adapt to unexpected issues in study execution or data that affect planned analyses. These revisions will be based on blinded review of the study and data.

#### 2 Investigational Plan

#### 2.1 Study design

This will be a multicenter, open-label, controlled study with two treatment arms running in parallel. A total of 188 patients of both genders and older than 18 years with type 2 diabetes and documented high cardiovascular risk and low grade inflammation will be randomly assigned to one of two treatment groups:

Arm A: treatment group: Rivaroxaban (5 mg b.i.d for the duration of 20 weeks, 52 weeks

duration for patients participating in the extension)

Arm B: control group: Aspirin (100 mg q.d. for the duration of 20 weeks, 52 weeks

duration for patients participating in the extension)



Figure 1: Trial overview

#### 2.2 Visit schedule

7 visits will be performed during the study. Visits will take place at week -2 (screening - V0), day 0 (randomization/baseline - V1), at week 2 (V2), 4 (V3), 8 (V4), 12 (safety/compliance - V5) and week 20 (end of treatment for the first study period with vascular function test - V6).

Additionally, 80 patients of the study population will perform 7 additional visits during the extension period. These visits will start after week 20. Patients attending the extension period performed a total of 14 study visits. The additional visits will take place at week 24 (V7), week 28 (V8), week 32 (V9), week 36 (V10), week 40 (V11), week 44 (V12) and week 52 (end of treatment extension - V13).

| VISIT | VO | V1 | V2 | V3 (TV) | V4 | V5 (TV) | V6 |
|---|---|---|---|---|---|---|---|
| WEEK | day -28 | day 0<br>(+/- 4 d) | 2<br>(+/- 2 d) | 4<br>(+/- 2 d) | 8<br>(+/- 2 d) | 12<br>(+/- 2 d) | 20<br>(+/- 2 d) |
| | SCREEN | BASELINE | TREAT | TREAT | TREAT | TREAT | EOT |
| STUDY INFORMED CONSENT | ✓ | | | | | | <b>√</b> A |
| SCREENING OF INCLUSION AND EXCLUSION CRITERIA | <b>*</b> | | | | | | |
| VITAL SIGNS (RADIAL PULSE,<br>BLOOD PRESSURE) | <b>√</b> | ~ | <b>~</b> | | ✓ | | <b>~</b> |
| RANDOMIZATION* | ✓ | | | | | | |
| BODY HEIGHT | <b>✓</b> | | | | | | |
| WAIST/HIP CIRCUMFERENCE<br>BODY WEIGHT | 1 | | | | | | 1 |
| ECG | ✓ | | | | | | |
| MEDICAL HISTORY | ✓ | | | | | | |
| CONCOMITANT MEDICATION/<br>ACUTE DISEASES | 1 | 1 | 1 | ~ | 4 | ~ | 1 |
| ARTERIAL STIFFNESS | | <b>✓</b> | | | | | ✓ |
| FOREARM BLOOD FLOW | | ✓ | | | | | ✓ |
| INFLAMMATION LABORATORY <sup>[1]</sup> | | <b>✓</b> | | | | | ✓ |
| SAFETY LABORATORY <sup>(3)</sup> | ✓ | ✓ | ✓ | | 4 | | ✓ |
| EFFICACY LABORATORY <sup>(2)</sup> | | <b>✓</b> | | | | | <b>~</b> |
| METABOLIC MARKER <sup>(4)</sup> | | 1 | | | | | 1 |
| SCREENING LABORATORY <sup>[5]</sup> | ✓ | | | | | | |
| CARDIOVASCULAR MARKER | | 1 | | | | | 1 |
| LDF INVESTIGATIONS | | <b>✓</b> | | | | | <b>4</b> |
| PLATELET ACTIVATION/<br>MITOGENIC POTENTIAL | | 1 | | | | | 1 |
| ADVERSE EVENT REPORTING | | ✓ | <b>*</b> | <b>√</b> | 4 | ✓ | ✓ |
| DISPENSING/RETURN OF<br>MEDICATION/<br>DRUG ACCOUNTABILITY | | ~ | <b>*</b> | | <b>*</b> | | ~ |
| PREGNANCY TEST | <b>√</b> | | | | | | |

Table 1: Study visits and parameters

| VISIT | V7 (TV) | V8 | V9 (TV) | V10 | V11 (TV) | V12 (TV) | V13 |
|---|---|---|---|---|---|---|---|
| WEEK | 24 | 28<br>(+/- 2 d) | 32<br>(+/- 2 d) | 36<br>(+/- 2 d) | 40 | 44<br>(+/- 2 d) | 52<br>(+/- 2 d) |
| | (+/- 2 d)<br>TREAT | TREAT | TREAT | TREAT | (+/- 2 d)<br>TREAT | TREAT | EOT<br>EXTEN-<br>SION |
| STUDY INFORMED CONSENT<br>FOR EXTENSION PERIOD | <b>*</b> | | | | | | |
| VITAL SIGNS (RADIAL PULSE,<br>BLOOD PRESSURE) | | <b>~</b> | | <b>*</b> | | | <b>*</b> |
| BODY HEIGHT | | | | | | | <b>~</b> |
| WAIST/HIP CIRCUMFERENCE<br>BODY WEIGHT | | | | | | | <b>*</b> |
| CONCOMITANT MEDICATION/<br>ACUTE DISEASES | > | * | <b>&gt;</b> | <b>&gt;</b> | > | > | <b>*</b> |
| ARTERIAL STIFFNESS | | | | | | | ✓ |
| FOREARM BLOOD FLOW | | | | | | | <b>*</b> |
| INFLAMMATION LABORATORY <sup>(1)</sup> | | | | | | | <b>√</b> |
| SAFETY LABORATORY <sup>(3)</sup> | | 4 | | <b>√</b> | | | <b>4</b> |
| EFFICACY LABORATORY <sup>(2)</sup> | | | | | | | <b>*</b> |
| METABOLIC MARKER <sup>(4)</sup> | | | | | | | <b>*</b> |
| LDF INVESTIGATIONS | | | | | | | <b>√</b> |
| ADVERSE EVENT REPORTING | ✓ | ✓ | ✓ | ✓ | ✓ | 4 | ✓ |
| DISPENSING/RETURN OF MEDICATION/ DRUG ACCOUNTABILITY | | <b>*</b> | | * | | | * |

Table 2: Study visits and parameters of extended treatment period

#### 2.3 Study objectives

Objectives of this clinical trial are the in vivo assessment of microvascular function using different non-invasive techniques and the in vitro assessment of biomarkers of endothelial damage, inflammation and coagulation/fibrinolysis before and after treatment with either aspirin or rivaroxaban in type 2 diabetic patients with high cardiovascular risk and inflammation. Furthermore possible functional interactions between mononuclear blood cells and platelets as well as expression of mRNA (and protein) within these cells before and after treatment in vitro will be assessed.

#### 2.3.1 Primary objectives

Primary objective is the difference of change of forearm blood flow with venous occlusion plethysmography at baseline and after forearm ischemia after 20 weeks treatment between rivaroxoban and aspirin therapy.

Additionally the difference of arterial stiffness after 52 weeks treatment (extension study) between rivaroxoban and aspirin therapy will be evaluated.

### 2.3.2 Secondary objectives

- Change of peripheral skin microcirculatory function (measured by Laser Doppler fluxometry;
   LDF) after 20 and 52 weeks of treatment
- LDF baseline
- LDF after ischemia (endothelial function)
- arterial stiffness measured by Mobilograph (IEM Inc.) after 20 weeks of treatment
- laboratory markers for endothelial function
- VCAM, ICAM, E-Selectin, ADMA, Nitrotyrosin, P-Selectin, CD40-L
- Microalbuminuria, eGFR
- composite of biomarkers of inflammation
- hsCRP, PAI-1, MCP-1, MMP-9, fibrinogen, leucocytes, MPO, IL-6, IL-8
- side effects: major bleeding according to ISTH, symptomatic thromboembolic events
- metabolic marker: HbA<sub>1c</sub>, lipids: triglycerides, LDL-C, HDL-C
- coagulation: von Willebrand-Factor, Fibrinogen, Prothrombinfragment 1 + 2, D-Dimer, Protein C, Protein S, TAT, Quick, aPTT
- cardiovascular marker: NT-proBNP, hs-Tnl, GDF-15, MR-ANP

Additional secondary objective for extension period:

• Difference of change of forearm blood flow with venous occlusion plethysmography at baseline and after forearm ischemia after 52 weeks treatment.

#### 2.3.3 Explorative study objective(s)

Assessment of platelet activation, measurement of mitogenic potential and risk benefit assessment.

#### 2.4 Sample size calculation

The first primary variable is the change of forearm blood flow with venous occlusion plethysmography ( $\Delta$ FBF) after forearm ischemia after 20 weeks of treatment. The sample size calculation is based on the following assumptions:

- Hypotheses: H0:  $\mu_{\Delta FBF, Riva} \leq \mu_{\Delta FBF, ASS}$ H1:  $\mu_{\Delta FBF, Riva} > \mu_{\Delta FBF, ASS}$
- Application of t-test for independent samples
- Type I error:  $\alpha = 0.05$
- Power: 1-ß = 0.90
- Estimated dropout rate: 25 %
- Minimum of expected clinical relevant difference between the groups in changes of maximal forearm blood flow ( $\Delta$ FBF) = 1.2 ml/100ml with an estimated standard deviation (STD)  $\sigma$  = 2.4 ml/100ml

Sample size should be at least N = 188 Patients (i.e. N/2 = 94 patients per arm) in order to achieve a valid number of 141 patients (per protocol analysis).

Additionally, the second primary variable is the difference of PWV between treatment groups at EOT Extension (after 52 week of treatment). The sample size calculation is based on the following assumptions:

H0: μ<sub>PWV, Riva</sub> = μ<sub>PWV, ASS</sub>

• H1:  $\mu_{PWV, Riva} \neq \mu_{PWV, ASS}$ 

• Type I error:  $\alpha = 0.05$ , t-test for independent samples

Power: 1-ß = 0.80

Estimated dropout rate: 20 %

• Minimum of expected clinical relevant difference between the groups in PWV = 0.7 m/s with an estimated standard deviation (STD) of  $\sigma$  = 1.0 m/s

Sample size should be N=80 patients (40 patients per arm) to achieve a valid number of 66 patients for per protocol analysis.

In summary the necessary sample size would be N=188 patients for the study up to week 20 including 80 patients for the extension up to week 52.

#### 3 Analysis Sets

For the analysis, patients not fulfilling the selection criteria of the trial ("all randomized") will be excluded from the statistical analysis. Only casuistic reports will be provided for this group.

#### 3.1 Full Analysis Set (FAS)

For the analysis, patients not fulfilling the selection criteria of the trial ("all randomized") will be excluded from the statistical analysis. Only casuistic reports will be provided for this group. All other patients will primarily be evaluated in an intent-to-treat analysis (ITT, FAS).

#### 3.2 Safety Analysis Set (SAF)

All patients having received at least one application of study medication are generally evaluable for safety and will be included in the safety analysis set.

#### 3.3 Per-Protocol Set (PPS)

Analyses of efficacy endpoints will be performed on the per protocol analysis set (PPS) defined as the subset of subjects of the FAS who have provided complete data of the target variable of interest at the first (V1) and last visit (V6/V13) and who have no major protocol deviations thought to impact the efficacy conclusions of the trial. The classification of protocol violation as major and minor will be done in a data review meeting that will take place after the database is clean.

#### 4 Analysis Variables

#### 4.1 Demographics

The following demographic characteristics will be summarized at baseline day 0: age (year), gender, race.

#### 4.2 Medical history

Information on following diagnostics will be recorded at baseline day 0: Pregnancy Test (done yes/no), result of pregnancy test (pregnant yes/no), ECG (yes/no), if "yes", ECG result ("normal", "minor findings", "major findings") Duration of diabetes
In- and exclusion criteria

#### 4.3 Concomitant medication and acute diseases

Medications taken will be recorded from the day of informed consent until the EOT visit (day 0-week 52). Patients who received a concomitant medication at any point of time will be counted in the category "yes". All patients who did not receive any concomitant medication in the course of the study will be counted in the category "no".

#### 4.4 Drug administration

The drug amount dispensed and returned will be recorded. Compliance (proportion of drug taken compared to drug dispensed) will be monitored.

#### 4.5 Efficacy Variables

Efficacy variables will be measured at day 0, weeks 20 and week 52:

Forearm blood flow (FBF) (mL/100mL): IR baseline, IR post-ischemic, IR post-ischemic (AUC)

#### Extension:

Arterial stiffness measured by pulse wave analysis: Pulse wave velocity (m/s), index of augmentation (%), peripheric and central blood pressure systolic/diastolic (mmHg)

Skin blood flow (measured by Laser Doppler):

Depth pre-ischemic blood flow (U), depth post-ischemic blood flow (U), shallow pre-ischemic blood flow (U) and shallow post-ischemic blood flow (U)

#### 4.6 Laboratory Variables

Several categories of laboratory variables are assessed:

- screening laboratory (day -28):
  hemoglobin, hematocrit, ALAT, ASAT, creatinine (PAP method), blood cell count (leucocytes, erythrocytes, platelets), total bilirubin, sodium, potassium, eGFR, HDL-C, triglycerides, cholesterine, urinary albumin/creatinin ratio, creatinine urine, hsCRP (if not available before screening visit according to in- and exclusion criteria), PAI1 (optional), urine pregnancy test
- inflammation laboratory (day 0, weeks 20, 52): hsCRP, PAI-1, MCP-1, MPO, IL-6, IL-8, MMP-9, fibrinogen
- efficacy laboratory for endothelial function and coagulation (day 0, weeks 20, 52):
   VCAM-1, ICAM-1, E-Selectin, P-Selectin, CD40L, von Willebrand factor, ADMA, nitrotyrosin, urinary albumin/creatinin ratio, eGFR, UACR, creatinin (serum), fibrinogen (immunolog), prothrombin fragment 1 and 2, TAT, D-Dimer, protein C, protein S, Quick, aPTT
- metabolic markers (day 0 (if not available, using of values at screening visit), weeks 20, 52):
   HbA<sub>1c</sub>, triglycerides, LDL-C, HDL-C, total cholesterine
- cardiovascular markers: NT-proBNP, hs-Tnl, GDF-15, MR-ANP
- bioassay data (subpopulation at day 0 and week 20): Thrombocytic micro-particles, vasodilatorstimulated phoshoprotein (VASP), serine-positive thrombocytes und thrombocyte proliferation rate.

#### 4.7 Safety Variables

#### 4.7.1 Vital Signs

Vital Signs will be collected in terms of:

Height (cm) (day 0, week 52)

Weight (kg), BMI (kg/m2), Waist and Hip circumference (cm) (day 0, weeks 2, 8, 20, 28, 36, 52) Radial pulse (bpm), systolic/diastolic blood pressure (mmHg) (day 0, weeks 2, 8, 20, 28, 36, 52)

#### 4.7.2 Safety laboratory

Safety laboratory variables will be monitored (day 0, weeks 2, 8, 20, 28, 36, 52): hemoglobin, hematocrit, ALAT, ASAT, creatinine (PAP method), blood cell count (leucocytes, erythrocytes, platelets), total bilirubin, sodium, potassium, eGFR

#### 4.7.3 Adverse Events and Serious Adverse Events

Adverse events and serious adverse events will be collected from first intake of study medication and then at each visit until the end of the study (day 0-week 52).

Bleedings (yes/no). If "yes" bleeding is classified as:

- major bleeding ("major")
- clinically relevant non-major bleeding ("CRNM")

Patients with major bleeding at any time in the course of the study will be counted in the category "major". All patients with CRNM but never "major" at any time will be counted in the category "CRNM". Only patients with minor bleedings but never CRNM are counted in the category "minor".

#### Adverse events:

All AE/SAE will be assessed and documented by the investigator according to the categories detailed below.

- Seriousness (yes/no):
  - Patients with SAE at any time in the course of the study will be counted in the category SAE. All patients with AE but not serious at any time will be counted in the category AE.
- Intensity (mild, moderate, severe)
- Causal relationship (yes/no)
- Action taken with study treatment (drug withdrawn, drug interrupted, dose reduced, dose not changed, dose increased, not applicable, unknown)
- Other specific treatments (none, remedial drug therapy, other)
- Outcome (recovered/resolved, recovered/resolved with sequelae, not recovered/not resolved, life-threatening, fatal, unknown)

#### 4.8 Definition of derived variables

#### 4.8.1 Primary variable

#### ΔFBF:

 $\Delta$ FBF (ml/100ml) will be composed of 5 IR baseline measurements and 8 measurements of post-ischemic blood flow. Repeated measurements for IR baseline per visit will be summarized by arithmetic mean.

Changes in FBF (ml/100ml) will be calculated as IR post-ischemic – IR baseline (mean).

#### 4.8.2 Secondary variables

Skin blood flow (LDF):

 $\Delta$  Depth: post-ischemic blood flow (depth) – pre-ischemic blood flow (depth)  $\Delta$  Shallow: post-ischemic blood flow (shallow) – pre-ischemic blood flow (shallow)

#### 5 Efficacy Endpoints

#### 5.1 Primary endpoint

Comparison of treatment groups for ΔFBF at week 20

Additional primary variable for extension period:

Comparison of treatment groups for pulse wave velocity at week 52

#### 5.2 Secondary endpoints

- Comparisons of groups and changes from baseline per treatment group for the following variables:
  - o PWV at week 52
  - o Maximal difference between baseline and post-ischemic skin blood flow FBF
  - Change of area under the FBF curve over 10 cycles of venous congestion (compared to baseline/day 0) at week 20 and EoT extension
  - Index of augmentation at weeks 20 and 52
  - o pulse wave velocity at 20 weeks and EoT Extension compared to baseline
  - o change of maximal postischemic forearm blood flow during reactive hyperaemia after 5 min of forearm ischemia (FBF max. ml/100ml) at EOT after 52 weeks (EOT Extension)
  - o laboratory parameters (see above) at weeks 20 and 52

#### 6 Statistical Methods

#### 6.1 Data Handling

Concentrations below the lower limit of quantification will be set to zero by laboratory. In case a set of continuous data contains zeros, an analysis in log scale (as described in 6.3) will be omitted.

#### 6.2 Descriptive or summary statistics

All continuous variables will be summarized by treatment group using the following statistics: n (non-missing sample size), number of missing values (Missing), arithmetic mean (Mean), standard deviation, (STD), median (Median), maximum (Max) and minimum (Min).

Tables for original (untransformed) data will be provided as well as tables for differences from baseline by visit. Boxplots will be presented for illustration.

For nominal or categorical data, frequencies and percentages (based on the non-missing sample size) will be tabulated for each category.

#### 6.3 Hypothesis Testing

Unless otherwise specified all hypotheses will be tested at a 5% level of significance against two-sided alternative hypotheses.

Continuous variables will be analyzed by the following test procedures:

First of all the assumption of normally distributed data will be checked with Shapiro-Wilk test by treatment group. If the hypothesis of normally distributed data cannot be rejected for both treatment groups treatments will be compared by an ANCOVA procedure which includes "treatment" as the main factor and "baseline value" as covariate. T-Tests for independent samples will be used to compare groups at baseline.

In the event that the normality assumption is not warranted, data will be log-transformed and normality assumption of the transformed data will be checked by Shapiro-Wilk test. In case of non-rejection of the hypothesis of normally distributed data for both treatment groups, ANCOVA procedure and t-tests as described above will be performed on the basis of log-transformed data.

Point estimates and 95% CI of the difference in (adjusted) mean change from baseline will be provided if data are evaluated on basis of an ANCOVA procedure.

Otherwise Mann-Whitney's-U test on the basis of original data will be applied for comparison of groups at baseline. Mann-Whitney's-U test on the basis of intra-individual differences to baseline will be applied for treatment comparison per visits after baseline. Wilcoxon's signed rank test will be applied to evaluate changes from baseline per treatment group.

Categorical variables with 2 categories will be analyzed using Fisher's exact test (with Yates correction) to compare proportions between treatment groups. Variables with more than 2 categories will be compared by Pearson's Chi-square test. Additionally for each category, the proportions of treatment groups are compared using an (asymptotic) z test. Significant differences in proportions will be flagged, p-values for the z-test will not be shown.

Missing values will not be imputed.

If necessary, modifications of this general procedure will be described in the following sections of chapter 6.

#### 6.4 Subject Disposition

Subject disposition analyses will be based on all enrolled subjects. The following summaries will be provided:

• Subject disposition, as the number of subjects screened, randomized and completed treatment will be summarized.

The following listings will be provided:

- Listing of subjects withdrawn or dropped out: date of baseline visit, date of the last visit, discontinued by reason
- If there are any protocol deviations, including violation of inclusion/exclusion criteria, and postenrollment deviations which will impact assessment of efficacy and safety endpoints, a listing will be generated.

#### 6.5 Demographics

Demographic characteristics will be summarized in total and by treatment groups (and center) on the basis of FAS, PPS and SAF. Listings of demographic characteristics will be presented.

#### 6.6 Medical History

Medical history will be summarized for FAS, PPS and SAF by each treatment group. Frequency tables will be provided for pregnancy test and ECG results.

#### 6.7 Concomitant medication and Acute Diseases

Medications taken will be recorded from the day of informed consent until the EOT visit (day 0-week 52). Patients who received a concomitant medication at any point of time will be counted in the category "yes". All patient who did not receive any concomitant medication in the course of the study will be counted in the category "no". Number and proportion of subjects taking prior/concomitant medication will be summarized.

#### 6.8 Compliance

The overall treatment compliance will be calculated as: [1- (overall amount of drug dispensed – overall amount of drug returned) / (overall amount of drug dispensed)]x 100%.

In addition to the overall compliance, the treatment compliance will be presented by the following specific ranges for each treatment group: <50%, <80%. Analysis of compliance will be based on FAS.

#### 6.9 Treatment exposure and observation period

The duration of treatment exposure period during the study is calculated as:

(last drug administration date – first drug administration date) + number of days to next visit after last drug administration.

The duration of observation period during the study is calculated as:

last contact date - randomization date +1.

The duration of exposure and the duration of observation period will be summarized for each treatment group (FAS, PPS and SAF).

#### 6.10 Analysis of baseline characteristics

Baseline data including demographics, anamnestic data, vital signs and laboratory values will be summarized by treatment group. Analyses will be repeated in SAF, FAS and PPS.

#### 6.11 Analysis of Efficacy Endpoints

All efficacy endpoints will be assessed for FAS, PPS and SAF.

#### 6.11.1 Analysis of Primary Endpoint

Primary study endpoint:

The hypothesis H0 is tested against the one-sided alternative hypothesis H1

```
H0: \mu_{\Delta FBF,Riva, week 20} \leq \mu_{\Delta FBF, ASS, week 20} vs. H1: \mu_{\Delta FBF, Riva, week 20} > \mu_{\Delta FBF, ASS, week 20}
```

by test procedures for continuous data. In case of non-rejection of the normality hypothesis an ANCOVA procedure for repeated measurements will be applied. For repeated measurements per subject an AR(1)-covariance-structure will be specified. Otherwise ANCOVA for repeated measurements will be based on (Blom-transformed) rank data.

Primary endpoint for the extension period:

The hypotheses

```
H0: \mu_{PWV, Riva, week 52} = \mu_{PWV, ASS, week 52} VS. H1: \mu_{PWV, Riva, week 52} \neq \mu_{PWV, ASS, week 52}
```

will be tested by procedure for continuous data.

Age, gender and duration of diabetes might represent confounding factors and could thus be included as covariates in the statistical model. Models incorporating different combinations of covariates are compared with respect to their model fit. The best fitting model according to the QIC (Quasi-Likelihood information) -criterion will be finally chosen for analysis.

Correction procedures for multiple comparisons are not necessary due to the fact that both primary endpoints consist in single comparisons addressing different variables.

#### 6.11.2 Analysis of Secondary Endpoints

All secondary endpoints will be analyzed according to the procedure for continuous variables. Correlations (original data and changes from baseline) might be calculated.

#### 6.12 Analysis of Safety Data

The summary of safety will be performed based on the SAF.

#### 6.12.1 Vital Signs

Summaries of vital sign variables will include original data and change from baseline by visit.

Blood pressure will be analyzed only by PWA because these measurements are regarded as more precise.

#### **6.12.2 Safety Laboratory Measurements**

Summaries of safety laboratory variables will include:

- Descriptive statistics of original values and differences from baseline
- The number (n) and percentage (%) of subjects with CSVs during study, depending on data.

#### **6.12.3** Adverse Events

Individual listings of treatment-emergent adverse events will be generated. The incidence of treatment-emergent adverse events, respectively, will be summarized using WHO SOC terms. Analysis of adverse events will be based on the SAF.

Listings of AEs, SAEs, ADRs and SADRs will be generated. The following variables will be included in the listing:

- Patient ID
- Treatment group
- Age/gender/race
- Verbatim Term
- AE start date and end date/ongoing
- AE Duration
- Study day onset
- Intensity
- Relationship of AE to study drug: unrelated or related
- Action taken
- Treatment
- Outcome

Listing of SADRs resulting in death and study discontinuation will also be generated.

#### 6.12.4 Bleedings

The results for major, CRNM, minor and total bleeding will be documented. Total bleeding includes any bleeding event (including CRNM, minor and major bleeding). These analyses will be performed on SAF and PPS.

#### 6.13 Interim analysis

Interim analyses are not planned.

#### 6.14 Reporting conventions

P-values  $\geq$  0.001 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "< 0.001". The mean, standard deviation and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles, such as median, or min and max will use the same number of decimal places as the original data. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 digits.

7 Appendix: Mock-Up tables, figures and listings

## 7.1 Subjects Disposition

| | Frequencies | | | | | |
|---|---|---|---|---|---|---|
| Patients | To | Total | | oxaban | Aspirin | |
| | N | % | N | % | N | % |
| Enrolled | | | | | | |
| Screening failures | | | | | | |
| Randomized | | | | | | |
| Study drug never administered | | | | | | |
| Treated | | | | | | |
| Did not complete study | | | | | | |
| Completed study | | | | | | |

| | Frequencies | | | | | |
|--------------|-------------|------|-------|--------|----|-------|
| Analysis Set | To | otal | Rivar | oxaban | As | pirin |
| | N | % | N | % | N | % |
| FAS | | | | | | |
| SAF | | | | | | |
| PPS | | | | | | |

| Exclusions | Frequencies | | | | | |
|------------|-------------------|---|---|---|---------|---|
| EXCIUSIONS | Total Rivaroxaban | | | | Aspirin | |
| from | N | % | N | % | N | % |
| FAS | | | | | | |
| SAF | | | | | | |
| PPS | | | | | | |

| December 5 colories from 546 | Frequencies | | | | | |
|---|---|---|---|---|---|---|
| Reasons for Exclusion from FAS (Screening Failures) | To | otal | Rivar | oxaban | Aspirin | |
| (Screening randles) | N | % | N | % | N | % |
| Study drug never administered | | | | | | |
| (all screening failures) | | | | | | |
| Study drug never administered | | | | | | |
| Non-Compliance | | | | | | |
| Data not complete | | | | | | |

| | Frequencies | | | | | |
|---|---|---|---|---|---|---|
| Reasons for Exclusion from SAF | Total | | Rivaroxaban | | Aspirin | |
| | N | % | N | % | N | % |
| Screening Failure | | | | | | |
| Study drug never administered | | | | | | |
| further reasons | | | | | | |

| | Frequencies | | | | | |
|---|---|---|---|---|---|---|
| Reasons for Exclusion from PPS | To | Total | | oxaban | Aspirin | |
| | N | % | N | % | N | % |
| Screening Failure | | | | | | |
| Study drug never administered | | | | | | |
| Non-Compliance | | | | | | |
| Withdrawal of consent | | | | | | |
| Study drug never administered | | | | | | |
| Data not complete | | | | | | |
| further reasons | | | | | | |

## 7.2 Demographics

| | | | | Freque | encies | | | Hypothesis Testing |
|---|---|---|---|---|---|---|---|---|
| Demog | raphics | Total | | Rivar | oxaban | As | pirin | Comparison of<br>Proportions |
| Variable | Category | N | % | N | % | N | % | p-Value |
| Gender | Female | | | | | | | |
| Gender | Male | | | | | | | |
| | European | | | | | | | |
| Dana | Asian | | | | | | | |
| Race | | | | | | | | |

| Demogr | aphics | | | | | | Origi | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Desc | criptive Sta | tistics | | | Normality | Comparis | on of Groups | at Baseline |
| Variable | Treatment | N | Missing | Mean | Median | STD | Max | p-Value | Effect | p-Value | 95% CI | |
| | Rivaroxaban | | | | | | | | | | | |
| Age | Aspirin | | | | | | | | | | | |
| | Total | | | | | | | - | - | - | - | |

7.3 Medical History

### 7.3.1 Medical History

| Duration of Diabetes | | | Origir | al Data |
|---|---|---|---|---|
| Duration of Diabetes | Descriptive Statistics Normality Comparison of Groups | | | |
| Treatment | N | N Missing Mean Median STD Min Max p-Value Effect p-Value 95% C | | |
| Rivaroxaban | | | | |
| Aspirin | | | | |

### 7.3.2 Concomitant medication

| Conconsitent | | | Frequ | iencies | | | Comparison of |
|---|---|---|---|---|---|---|---|
| Concomitant medication | To | otal | Rivaro | xaban | As | pirin | Proportions |
| medication | N | % | N | % | N | % | p-Value |
| yes | | | | | | | |
| no | | | | | | | |

### 7.3.3 ECG and Pregnancy Test

| | Λ. | Andical History | | | Freque | encies | | |
|---|---|---|---|---|---|---|---|---|
| | IV | 1edical History | To | otal | Rivar | oxaban | As | pirin |
| Variable | | Category | N | % | N | % | N | % |
| | | Normal | | | | | | |
| | | Abnormal, clinically not significant | | | | | | |
| ECG | yes | Abnormal, clinically significant | | | | | | |
| | | total | | | | | | |
| | no | | | | | | | |
| Pregnancy yes | | | | | | | | |
| test done | no | | | | | | | |

## 7.4 Compliance

| Caman | lianaa [0/] | | | | | | Origin | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Comp | liance [%] | | | Desc | riptive Stati | stics | | | Normality | Con | nparison of G | roups |
| Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| Wook 2 | Rivaroxaban | | | | | | | | | | | |
| Week 2 | Aspirin | | | | | | | | | | | |
| Week 4 | Rivaroxaban | | | | | | | | | | | |
| vveek 4 | Aspirin | | | | | | | | | | | |
| Week 8 | Rivaroxaban | | | | | | | | | | | |
| vveek o | Aspirin | | | | | | | | | | | |
| Week 20 | Rivaroxaban | | | | | | | | | | | |
| Week 20 | Aspirin | | | | | | | | | | | |
| Week 28 | Rivaroxaban | | | | | | | | | | | |
| WEEK 20 | Aspirin | | | | | | | | | | | |
| Week 36 | Rivaroxaban | | | | | | | | | | | |
| Week 30 | Aspirin | | | | | | | | | | | |
| Week 52 | Rivaroxaban | | | · | | · | | | | | | |
| WEEK 32 | Aspirin | | | | | | | | | | | |
| Overall | Rivaroxaban | | | | | | | | | | | |
| Overall | Aspirin | | | | | | | | | | | |

| | | | Fı | requencies | | | Comparison of |
|---|---|---|---|---|---|---|---|
| Total Compliance | Total | | Riva | aroxaban | Α | spirin | Proportions |
| | N | % | N | % | N | % | p-Value |
| < 50% | | | | | | | |
| ≥ 50% and < 80% | | | | | | | |
| ≥ 80% | | | | | | | |

## 7.5 Treatment exposure and observation period

| Durg | ation | | | | | | Origir | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dura | ation | | | Desc | riptive Stat | istics | | | Normality | Con | nparison of G | iroups |
| | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| Treatment | Rivaroxaban | | | | | | | | | | | |
| exposure | Aspirin | | | | | | | | | | | |
| Observation | Rivaroxaban | | | • | | | | | | | | |
| period | Aspirin | | | | | | | | | | | |

## 7.6 Efficacy Endpoints

## 7.6.1 Forearm Blood Flow (FBF)

| | | FBF | | | | | | | Origin | al Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | LRL | | | | Desc | riptive Stati | stics | | | Normality | Compariso | on of Groups | at Baseline |
| Variable | Visit | Value | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| A EDE | | Post1- | Rivaroxaban | | | | | | | | | | | |
| ΔFBF | | baseline | Aspirin | | | | | | | | | | | |
| | | Post2- | Rivaroxaban | | | | | | | | | | | |
| | | baseline | Aspirin | | | | | | | | | | | |
| | | Post3- | Rivaroxaban | | | | | | | | | | | |
| | | baseline | Aspirin | | | | | | | | | | | |
| | | Post4- | Rivaroxaban | | | | | | | | | | | |
| | Day 0 | baseline<br>Post5- | Aspirin | | | | | | | | | | | |
| | Day 0 | | Rivaroxaban | | | | | | | | | | | |
| | | baseline | Aspirin | | | | | | | | | | | |
| | | Post6- | Rivaroxaban | | | | | | | | | | | |
| | | baseline | Aspirin | | | | | | | | | | | |
| | | Post7- | Rivaroxaban | | | | | | | | | | | |
| | | baseline | Aspirin | | | | | | | | | | | |
| | | Post8- | Rivaroxaban | | | | | | | | | | | |
| | | baseline | Aspirin | | | | | | | | | | | |
| | Week | | Rivaroxaban | | | | | | | | | | | |
| | 20 | | Aspirin | | | | | | | | | | | |
| | Week | | Rivaroxaban | | | | | | | | | | | |
| | 52 | | Aspirin | | | | | | | | | | | |

| | FBF | | | | | Origin | al Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | FBF | | Desci | riptive Stat | istics | | | Normality | Comparis | on of Group: | s at Baseline |
| D.4-11 | Max Day 0 | | | | | | | | | | |
| IR post- | Max. Day 0 Aspirin | | | | | | | | | | |
| ischemic | Week 20 | Rivaroxaban | | | | | | | | | |

#### MicroVasc-DIVA

| | | Aspirin | |
|----------------------|----------|-------------|---|
| | Week 52 | Rivaroxaban | |
| | week 52 | Aspirin | |
| ID post | Day 0 | | · |
| IR post-<br>ischemic | Day 0 | | |
| ischemic<br>(AUC) | Week 20 | | |
| | vveek 20 | | |
| | Week 52 | | · |
| | Week 32 | | · |

| | ΔFBF | | | | | | | Chang | es from | Baseline | Day 0 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (Di | ifferenzen zı | ı V0) | | | De | escriptive Stat | istics | | | Com | parison to E | Baseline | Com | oarison of ( | Groups |
| Visit | Value | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| Week 20 | Post1- | Rivaroxaban | | | | | | | | | | | | | |
| Week 20 | baseline | Aspirin | | | | | | | | | | | | | |
| | Post2- | Rivaroxaban | | | | | | | | | | | | | |
| | baseline | Aspirin | | | | | | | | | | | | | |
| | Post3- | Rivaroxaban | | | | | | | | | | | | | |
| | baseline | Aspirin | | | | | | | | | | | | | |
| | Post4- | Rivaroxaban | | | | | | | | | | | | | |
| | baseline | Aspirin | | | | | | | | | | | | | |
| | Post5- | Rivaroxaban | | | | | | | | | | | | | |
| | baseline | Aspirin | | | | | | | | | | | | | |
| | Post6- | Rivaroxaban | | | | | | | | | | | | | |
| | baseline | Aspirin | | | | | | | | | | | | | |
| | Post7- | Rivaroxaban | | | | | | | | | | | | | |
| | baseline | Aspirin | | | | | | | | | | | | | |
| | Post8- | Rivaroxaban | | | | | | | | | | | | | |
| | Post8-<br>baseline | l — | Aspirin | | | | | | | | | | | | |

| | | | | | | | | Chang | es from | Baseline | Day 0 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | FBF | | | | De | escriptive Stat | istics | | | Com | nparison to E | Baseline | Comp | oarison of ( | Groups |
| Variable | Visit | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| Mari | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Max.<br>IR post- | Week 20 | Aspirin | | | | | | | | | | | | | |
| ischemic | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | WEEK 32 | Aspirin | | | | | | | | | | | | | |
| | Week 20 | | | | | | | | | | | | | | |
| IR post-<br>ischemic | WEEK 20 | | | | | | | | | | | | | | |
| (AUC) | Week 52 | | | | | | | | | | | | | | |
| | VVEEK JZ | | | | | | | | | | | | | | |

### 7.6.2 Pulse Wave Analysis

| | PWA | | | | | | | Origir | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | PVVA | | | | Desc | riptive Stat | istics | | | Normality | Comparis | on of Groups | at Baseline |
| Variable | Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| Dules Marie | Day 0 | Rivaroxaban | | | | | | | | | | | |
| Pulse Wave<br>Velocity | Day 0 | Aspirin | | | | | | | | | | | |
| (m/s) <sup>*</sup> | Week 20 | Rivaroxaban | | | | | | | | | | | |
| | week 20 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | week 52 | Aspirin | | | | | | | | | | | |
| leden of | Day 0 | Rivaroxaban | | | | | | | | | | | |
| Index of Augmentation | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | | | |
| | Week 20 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | week 32 | Aspirin | | | | | | | | | | | |
| | Day 0 | Rivaroxaban | | | | | | | | | | | |

#### MicroVasc-DIVA

| Peripheral | | Aspirin |
|----------------------------|----------|-------------|
| Systolic Blood<br>Pressure | Wash 20 | Rivaroxaban |
| | Week 20 | Aspirin |
| | Week 52 | Rivaroxaban |
| | Week 32 | Aspirin |
| Dorinhoral | Day 0 | Rivaroxaban |
| Peripheral<br>Diastolic | Day 0 | Aspirin |
| Blood | Week 20 | Rivaroxaban |
| Pressure | Week 20 | Aspirin |
| | Week 52 | Rivaroxaban |
| | VVEEK 32 | Aspirin |
| Central | Day 0 | Rivaroxaban |
| Systolic Blood | Dayo | Aspirin |
| Pressure | Week 20 | Rivaroxaban |
| | WCCK 20 | Aspirin |
| | Week 52 | Rivaroxaban |
| | WCCK 32 | Aspirin |
| Central | Day 0 | Rivaroxaban |
| Diastolic | Day 0 | Aspirin |
| Blood<br>Pressure | Week 20 | Rivaroxaban |
| FIESSUIE | | Aspirin |
| | Week 52 | Rivaroxaban |
| | .vcck 32 | Aspirin |

| | | | | | | | | Chang | es from | Baseline | Day 0 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | PWA | | | | De | escriptive Stat | istics | | | Com | parison to E | Baseline | Com | parison of ( | Groups |
| Variable | Visit | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| Pulse | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Wave | Week 20 | Aspirin | | | | | | | | | | | | | |
| Velocity | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| (m/s) | Week 32 | Aspirin | | | | | | | | | | | | | |
| Index of | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Augmenta- | Week 20 | Aspirin | | | | | | | | | | | | | |
| tion | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | week 52 | Aspirin | | | | | | | | | | | | | |
| Darinharal | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Peripheral<br>Systolic | Week 20 | Aspirin | | | | | | | | | | | | | |
| Blood | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| Pressure | WEEK 32 | Aspirin | | | | | | | | | | | | | |
| Peripheral | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Diastolic | WEEK 20 | Aspirin | | | | | | | | | | | | | |
| Blood | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| Pressure | Week 32 | Aspirin | | | | | | | | | | | | | |
| Central | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Systolic | Week 20 | Aspirin | | | | | | | | | | | | | |
| Blood | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| Pressure | week 52 | Aspirin | | | | | | | | | | | | | |
| | )M/a al. 20 | Rivaroxaban | | | | | | | | | | | | | |
| Central<br>Diastolic | Week 20 | Aspirin | | | | | | | | | | | | | |
| Blood | M/ 52 | Rivaroxaban | | | | | | | | | | | | | |
| Pressure | Week 52 | Aspirin | | | | _ | | | | | | | | | |

## 7.6.3 Laser Doppler fluxometry (LDF)

| | LDF | | | | | | | Origin | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | LDF | | | | Desc | criptive Stat | istics | | | Normality | Comparis | on of Groups | at Baseline |
| Variable | Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| A Double | Day 0 | Rivaroxaban | | | | | | | | | | | |
| Δ Depth | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | | | |
| | Week 20 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | Week 32 | Aspirin | | | | | | | | | | | |
| Δ Shallow | Day 0 | Rivaroxaban | | | | | | | | | | | |
| Δ Shallow | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | | | |
| | Week 20 | Aspirin | | | | | | | | | | | |
| | Mook F2 | Rivaroxaban | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | |

| | | | | | | | | Chang | es from | Baseline | Day 0 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | LDF | | | | De | escriptive Stat | istics | | | Com | parison to B | aseline | Comp | oarison of C | Groups |
| Variable | Visit | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| A Donth | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Δ Depth | Week 20 | Aspirin | | | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 32 | Aspirin | | | | | | | | | | | | | |
| Δ Shallow | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Δ Shallow | Week 20 | Aspirin | | | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 32 | Aspirin | | | | | | | | | | | | | |

## 7.7 Efficacy Laboratory

### 7.7.1 Inflammation Laboratory

| Inflan | nmation Labo | ratory | | | | | | Origir | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| IIIIIdII | IIIIIaliOII LabC | iratory | | | Desc | riptive Stati | stics | | | Normality | Comparis | on of Groups | at Baseline |
| Variable | Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| h-CDD | Day 0 | Rivaroxaban | | | | | | | | | | | |
| hsCRP | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | - | - | - |
| | vveek 20 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | vveek 52 | Aspirin | | | | | | | | | | | |
| DAL 4 | Day 0 | Rivaroxaban | | | | | | | | | | | |
| PAI-1 | Day 0 | Aspirin | | | | | | | | | | | |
| | W1-20 | Rivaroxaban | | | | | | | | | - | - | - |
| | Week 20 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | |
| | • | | • | | •• | further v | /ariables | • | • | | | • | |

| Inflan | omation Lab | oratory | | | | | | Chang | es from | Baseline | Day 0 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| IIIIIaii | nmation Lab | oratory | | | De | escriptive Stat | istics | | | Com | parison to B | aseline | Com | parison of G | roups |
| Variable | Changes | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| h.CDD | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| hsCRP | Week 20 | Aspirin | | | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | vveek 32 | Aspirin | | | | | | | | | | | | | |
| DAL 4 | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| PAI-1 | vveek 20 | Aspirin | | | | | | | | | | | | | |
| | Wash 52 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | | | |

..... further variables.....

### 7.7.2 Laboratory for Endothelian Function and Coagulation

| Efficacy La | boratory for | Endothelial | | | | | | Origir | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Funct | ion and Coag | ulation | | | Desc | riptive Stati | stics | | | Normality | Comparis | son of Groups | at Baseline |
| Variable | Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| V/CANA 1 | Day 0 | Rivaroxaban | | | | | | | | | | | |
| VCAM-1 | Day 0 | Aspirin | | | | | | | | | | | |
| | Maak 20 | Rivaroxaban | | | | | | | | | - | - | - |
| | Week 20 | Aspirin | | | | | | | | | | | |
| | Mook F2 | Rivaroxaban | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | |
| 10000 | Day 0 | Rivaroxaban | | | | | | | | | | | |
| ICAM-1 | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | - | - | - |
| | Week 20 | Aspirin | | | | | | | | | | | |
| | Mook E2 | Rivaroxaban | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | |
| | | | | | | further \ | /ariables | | | | | | |

| Efficacy La | boratory for | · Endothelial | | | | | | Chang | es from | Baseline | Day 0 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Funct | ion and Coag | gulation | | | De | escriptive Stat | istics | | | Com | parison to B | aseline | Com | parison of G | roups |
| Variable | Changes | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| VCAM-1 | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| VCAIVI-1 | Week 20 | Aspirin | | | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | week 52 | Aspirin | | | | | | | | | | | | | |
| ICAM-1 | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| ICAIVI-1 | week 20 | Aspirin | | | | | | | | | | | | | |
| | Wook F2 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | 1 | | |
| | | | | | | 1 | further varia | ables | | | | | • | | |

..... similar table for Metabolic Markers and bioassay data ......

## 7.8 Safety Variables

### 7.8.1 Vital Signs

| | Vital Signs | | | | | | | Origin | nal Data | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Vital Signs | | | | Desc | criptive Stati | stics | | | Normality | Comparis | son of Groups | at Baseline |
| Variable | Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | p-Value | Effect | p-Value | 95% CI |
| I I a lada k | Day 0 | Rivaroxaban | | | | | | | | | | | |
| Height | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | - | - | - |
| | Week 32 | Aspirin | | | | | | | | | | | |
| Weight | Day 0 | Rivaroxaban | | | | | | | | | | | |
| weight | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | - | - | - |
| | WEEK 20 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | VVEEK 32 | Aspirin | | | | | | | | | | | |
| Radial Pulse | Day 0 | Rivaroxaban | | | | | | | | | | | |
| Radiai Puise | Day 0 | Aspirin | | | | | | | | | | | |
| | Week 2 | Rivaroxaban | | | | | | | | | - | - | - |
| | VVCCK Z | Aspirin | | | | | | | | | | | |
| | Week 8 | Rivaroxaban | | | | | | | | | | | |
| | WCCKO | Aspirin | | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | | | | |
| | WCCK 20 | Aspirin | | | | | | | | | | | |
| | Week 28 | Rivaroxaban | | | | | | | | | | | |
| | WCCK 20 | Aspirin | | | | | | | | | | | |
| | Week 36 | Rivaroxaban | | | | | | | | | | | |
| | WCCK 30 | Aspirin | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | |
| | WCCR JZ | Aspirin | | | | | | | | | | | |
| | | | | | | further v | ariables | | | | | | |

| | Vital Ciana | | | | | | | Char | iges fron | n Baseline | e V1 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Vital Signs | | | | De | escriptive Stat | istics | | | Comp | parison to Ba | aseline | Com | parison of G | roups |
| Variable | Visit | Treatment | N | Missing | Mea<br>n | Median | STD | Min | Max | Effect | p-Value | 95% CI | Effect | p-Value | 95% CI |
| \\/a:=b+ | Week 20 | Rivaroxaban | | | | | | | | | | | | | |
| Weight | week 20 | Aspirin | | | | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | | | | |
| | week 52 | Aspirin | | | | | | | | | | | | | |
| Dedial | Week 2 | Rivaroxaban | | | | | | | | | | | | | |
| Radial<br>Pulse | vveek 2 | Aspirin | | | | | | | | | | | | | |
| | Wash 0 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 8 | Aspirin | | | | | | | | | | | | | |
| | Maak 20 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 20 | Aspirin | | | | | | | | | | | | | |
| | Week 28 | Rivaroxaban | | | | | | | | | | | | | |
| | week 28 | Aspirin | | | | | | | | | | | | | |
| | Maak 20 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 36 | Aspirin | | | | | | | | | | | | | |
| | Mook F2 | Rivaroxaban | | | | | | | | | | | | | |
| | Week 52 | Aspirin | | | | | | | | | | | | | |
| further va | ariables | | • | | | | • | • | | | | | | | |

### 7.8.2 Safety Laboratory

| Safety Laboratory | | | Original Data | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Descriptive Statistics | | | | | | | | Comparison of Groups | |
| Variable | Visit | Treatment | N | Missing | Mean | Median | STD | Min | Max | Effect | p-value | 95% CI |
| Hemoglobin | Day 0 | Rivaroxaban | | | | | | | | | | |
| | | Aspirin | | | | | | | | | | |
| | Week 2 | Rivaroxaban | | | | | | | | | | |
| | | Aspirin | | | | | | | | | | |
| | Week 8 | Rivaroxaban | | | | | | | | | | |
| | | Aspirin | | | | | | | | | | |
| | Week 20 | Rivaroxaban | | | | | | | | - | | |
| | | Aspirin | | | | | | | | | | |
| | Week 28 | Rivaroxaban | | | | | | | | | | |
| | | Aspirin | | | | | | | | | | |
| | Week 36 | Rivaroxaban | | | | | | | | _ | | |
| | | Aspirin | | | | | | | | | | |
| | Week 52 | Rivaroxaban | | | | | | | | | | |
| | | Aspirin | | | | | | | | | | |

| | | | | Comparison of | | | | |
|---|---|---|---|---|---|---|---|---|
| Safety Laboratory CSV's | | | Total | | Rivaroxaban | | spirin | Proportions* |
| | | N | % | N | % | N | % | p-Value |
| Total | Number of Patients | | | | | | | |
| Total | Number of Events | | | | | | | |
| Homoglobin | Number of Patients | | | | | | | |
| Hemoglobin | Number of Events | | | | | | | |
| | further variables | | | | | | | |

<sup>\*</sup>can only be calculated for number of patients

#### 7.8.3 Adverse Events

| | | | | Comparison of | | | | |
|---|---|---|---|---|---|---|---|---|
| Adverse Events | | | Total | | Rivaroxaban | | spirin | Proportions |
| | | N | % | N | % | Ν | % | p-Value |
| Number of | AE | | | | | | | |
| | SAE | | | | | | | |
| Patients | ADR | | | | | | | |
| | SADR | | | | | | | |
| | AE | | | | | | | - |
| Number of<br>Events | SAE | | | | | | | |
| | ADR | | | | | | | |
| | SADR | | | | | | | |

## 7.8.4 Bleedings

| | | | | Comparison of | | | | |
|---|---|---|---|---|---|---|---|---|
| Bleedings | | | Total | | Rivaroxaban | | spirin | Proportions |
| | | N | % | N | % | N | % | p-Value |
| | Major | | | | | | | |
| Number of | CRNM | | | | | | | |
| Patients | Minor | | | | | | | |
| | Total Bleeding | | | | | | | |
| | Major | | | | | | | - |
| Number of<br>Events | CRNM | | | | | | | |
| | Minor | | | | | | | |
| | Total Bleeding | | | | | | | - |